CLINICAL TRIAL: NCT07260994
Title: Comparative Effect of High-Level Versus Low-Level Laser Therapy on Nerve Root Function Among Healthy Young Adults: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taif A. M. Omran (Other)
Collaborators: University of Sharjah (Other)
Responsible Party: Sponsor-Investigator, Taif A. M. Omran, Master Student, University of Sharjah
Organization: University of Sharjah (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-25-06-24-03-PG
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study will be single-blind where the participants will be blinded to group assignments. While the primary investigator will be aware about the group assignment. Participants will be kept unaware about their group assignment, will be asked to complete a consent form explaining the study thoroughly, except the information related to the number of groups involved in the study, and will be provided by the additional information related to the group assignment after the completion of the study (Monaghan et al., 2021; Simon et al., 2021).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HILT group (Active Comparator): Participants in HILT group will receive laser therapy with a wavelength of 1064 nm, frequency of 25 Hz, output power of 7 W, and energy dose of 120 J/cm^2, intervention will be delivered through non-contact mode, by using the Zimmer MedizinSysteme device (OptonPro, Germany) to deliver high-intensity laser over C6, C7, and C8 nerve roots as they exit the spinal column.
  Interventions: Radiation: High-intensity laser therapy
- LLLT group (Active Comparator): Participants in LLLT group will receive laser therapy with wavelength of 905nm, frequency of 5 kHz output power of 25mW, and energy dose of 2 J/cm^2, intervention will be delivered through contact mode, by using the Enraf-Nonius Endolaser device (South Africa) to deliver low-level laser over C6, C7, and C8 nerve roots as the exit the spinal column.
  Interventions: Radiation: Low-level laser therapy
- Sham laser group (Sham Comparator): For the participants in the sham group, the same procedure will be followed, but with having the laser device turned off.
  Interventions: Radiation: Sham laser

INTERVENTIONS:
Radiation: High-intensity laser therapy — Participants in HILT group will receive laser therapy with a wavelength of 1064 nm, frequency of 25 Hz, output power of 7 W, and energy dose of 120 J/cm^2, intervention will be delivered through non-contact mode, by using the Zimmer MedizinSysteme device (OptonPro, Germany) to deliver high-intensity laser over C6, C7, and C8 nerve roots as they exit the spinal column.
  Arms: HILT group
Radiation: Low-level laser therapy — Participants in LLLT group will receive laser therapy with wavelength of 905nm, frequency of 5 kHz output power of 25mW, and energy dose of 2 J/cm^2, intervention will be delivered through contact mode, by using the Enraf-Nonius Endolaser device (South Africa) to deliver low-level laser over C6, C7, and C8 as they exit the spinal column.
  Arms: LLLT group
Radiation: Sham laser — For the participants in the sham group, the same procedure will be followed, but with having the laser device turned off.
  Arms: Sham laser group

SUMMARY:
Study title: Comparative Effect of High-Level Versus Low-Level Laser Therapy on Nerve Root Function Among Healthy Young Adults: A Randomized Controlled Trial You are invited to participate in a research study to investigate the short-term effect of high-intensity laser therapy (HILT), low-level laser therapy (LLLT), and sham laser on nerve root function among healthy adults.

Participation is entirely voluntary, and you may withdraw from the study at any time without penalty or need for justifications if you choose to do so.

What is the aim of the study? The objective of the current study is to investigate the short-term effect of high-intensity laser therapy (HILT), low-level laser therapy (LLLT), and sham laser on nerve root function among healthy adults.

Type of participants? We are recruiting participants aged 18-30 years of both genders without any musculoskeletal or neurological disorder involving the upper extremities, non-smokers, and if they expressed their wellness to participate in the current study.

What will participants be asked to do? The purpose of this study is to investigate the short-term effect of high-intensity laser therapy, low-level laser therapy, and sham laser on nerve root function among healthy adults.

If you agree to take part:

* First, we will check if you are eligible for the study.
* If you are eligible and give your consent, you will be randomly placed into one of three groups:

  1. High-intensity laser therapy group
  2. Low-level laser therapy group
  3. Sham (placebo) group - in this group, the laser device will look and feel the same, but it will not actually deliver laser treatment.
* If you are in the sham group, you will not receive active laser therapy. This is important for the scientific accuracy of the study, as it allows us to compare the effects of real laser therapy with no treatment. You will not know which group you are in during the study, but you will be informed after your participation is complete.
* You will attend 9 short sessions over 3 weeks (3 sessions per week). Each session will last about 5-10 minutes.
* To measure nerve function before laser application (Step 1):

  1. A small gel will be used to place two sensors on your head (these can be removed easily).
  2. Three nerves in your arm will be tested using very light, safe electrical pulses delivered through a small hand-held electrode held in place with a strap.
  3. This helps us measure how your nerves are working before laser treatment by measuring the peak-to-peak amplitude and latency of N20 point of the brain through analyzing the brain waves.
* Laser or sham application (Step 2):

  1. A researcher will apply the laser (or sham) to three spots on your neck.
  2. Each spot will receive laser for about 2 minutes.
  3. The laser used is safe, does not cause heat, and you will not feel any burning.
* Measuring nerve function again (Step 3):

The same nerve test from step 1 will be repeated to see if there are any changes after the laser application.

* Men do not need to remove any clothing.
* Women who wear a headscarf will be asked to temporarily remove it so the head sensors can be placed. This will be done in a private room by a female researcher only, with doors locked and separators used to ensure complete privacy.
* Male participants will also be attended to by a male researcher in the same respectful and private way.
* It is very important to note that you may be assigned to a group where the laser is not actually turned on (sham group). This is important for the scientific accuracy of the study.
* You will be told which group you were in after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals deemed to be eligible to participate in the current study if they aged between 18 and 30 years of both genders, without any musculoskeletal or neurological disorder involving the upper extremities, non-smokers, and if they expressed their wellness to participate in the current study.

Exclusion Criteria:

* Individuals will be excluded if they have a history of cervical spine disorders; significant cervical disc herniation, spinal narrowing, cervical nerve root compression, or cervical spinal cord dysfunction; a history of severe and frequent migraines, shoulder diseases, fibromyalgia, rheumatic or rheumatoid diseases, mental illnesses, severe osteoporosis, significant spinal deformities, or serious neurological, cardiovascular, or pulmonary conditions; the presence of fever, infection, tumors; cognitive or emotional disorders; or pregnant or nursing women (Xie et al., 2025).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
N20 peak-to-peak amplitude and latency | N20 peak-to-peak amplitude and latency of C6, 7, and C8 will be measured at baseline and immediately after laser therapy application.
  The main outcome measure used to assess the nerve root function will be the N20 peak-to-peak amplitude and latency by using the dermatomal somatosensory evoked potentials (DSEPs).

CONTACTS AND LOCATIONS:
Overall Officials: Taif Omran, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates